CLINICAL TRIAL: NCT02242682
Title: Video Education: Capitalizing on Caregiver Time Spent in the Pediatric Emergency Department Waiting Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nina Muhammad, Pediatric Emergency Medicine Fellow, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 527345
Record Dates: First submitted 2014-09-02; First posted 2014-09-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Child Passenger Seat Safety

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): This group of subjects will not be exposed to a video during their time in the ED waiting room
- Child passenger safety video (Experimental): This group of subjects will be exposed to a video during their time in the ED waiting room
  Interventions: Other: Child passenger safety video

INTERVENTIONS:
Other: Child passenger safety video
  Arms: Child passenger safety video

SUMMARY:
The purpose of this study is to determine if video education is an effective means of caregiver education in the waiting room of a pediatric emergency department (ED). This will be tested with the showing of a child passenger safety video.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of patients presenting to Children's Hospital of Wisconsin for treatment
* family use of automobile for transportation

Exclusion Criteria:

* non-English speaking caregivers
* triage level 1 or 2 or requiring immediate medical attention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Efficacy: Difference in caregiver knowledge on a questionnaire | day 0 in the ED
  A knowledge questionnaire will be completed by caregivers in control and intervention groups

SECONDARY OUTCOMES:
Retention | up to 4 weeks after enrollment
  A knowledge questionnaire for caregivers will be given at phone follow up 4 weeks after initial enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Wheeler JG, Fair M, Simpson PM, Rowlands LA, Aitken ME, Jacobs RF. Impact of a waiting room videotape message on parent attitudes toward pediatric antibiotic use. Pediatrics. 2001 Sep;108(3):591-6. doi: 10.1542/peds.108.3.591. PMID 11533323
- [Background] Dunn RA, Shenouda PE, Martin DR, Schultz AJ. Videotape increases parent knowledge about poliovirus vaccines and choices of polio vaccination schedules. Pediatrics. 1998 Aug;102(2):e26. doi: 10.1542/peds.102.2.e26. PMID 9685472
- [Background] Macy ML, Davis MM, Clark SJ, Stanley RM. Parental health literacy and asthma education delivery during a visit to a community-based pediatric emergency department: a pilot study. Pediatr Emerg Care. 2011 Jun;27(6):469-74. doi: 10.1097/PEC.0b013e31821c98a8. PMID 21629152
- [Background] Shenoi R, Saz EU, Jones JL, Ma L, Yusuf S. An emergency department intervention to improve knowledge of child passenger safety. Pediatr Emerg Care. 2010 Dec;26(12):881-7. doi: 10.1097/PEC.0b013e3181fe909f. PMID 21088639
- [Background] Schnellinger M, Finkelstein M, Thygeson MV, Vander Velden H, Karpas A, Madhok M. Animated video vs pamphlet: comparing the success of educating parents about proper antibiotic use. Pediatrics. 2010 May;125(5):990-6. doi: 10.1542/peds.2009-2916. Epub 2010 Apr 12. PMID 20385634
- [Background] Uherick L, Gorelick MH, Biechler R, Brixey SN, Melzer-Lange M. Validation of two child passenger safety questionnaires. Inj Prev. 2010 Oct;16(5):343-7. doi: 10.1136/ip.2009.022681. Epub 2010 Aug 30. PMID 20805618
- [Background] Durbin DR, Elliott MR, Winston FK. Belt-positioning booster seats and reduction in risk of injury among children in vehicle crashes. JAMA. 2003 Jun 4;289(21):2835-40. doi: 10.1001/jama.289.21.2835. PMID 12783914
- See also: Related Info — http://www.chop.edu/service/car-seat-safety-for-kids/car-seat-safety-by-age/for-your-4-to-8-year-old-child.html